CLINICAL TRIAL: NCT00125359
Title: A Phase II Clinical Study of Erlotinib (Tarceva) and Bexarotene (Targretin) Oral Capsules in Patients With Advanced Non-small Cell Lung Cancer
Brief Title: Study of Tarceva and Targretin Oral Capsules in Patients With Advanced Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Konstantin Dragnev (Other)
Collaborators: Ligand Pharmaceuticals (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Konstantin Dragnev, Associate Professor of Medicine, Dartmouth-Hitchcock Medical Center
Organization: Dartmouth-Hitchcock Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D-0440
Record Dates: First submitted 2005-07-29; First posted 2005-08-01 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Carcinoma, Non-small-cell Lung
Keywords: tarceva; targretin; non-small cell lung cancer; Carcinoma, non-small cell lung cancer; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Carcinoma | interventions — Erlotinib Hydrochloride; Bexarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): All eligible patients will receive continuous daily oral erlotinib 150mg with daily bexarotene oral capsules 400mg.
  Interventions: Drug: erlotinib and bexarotene

INTERVENTIONS:
Drug: erlotinib and bexarotene — Daily Erlotinib 150mg and daily bexarotene oral capsules 400mg.

SUMMARY:
The purpose of this study is to learn about the effects of two new anticancer drugs, erlotinib (Tarceva) and bexarotene (Targretin), when treating patients with advanced lung cancer.

Erlotinib is approved by the Food and Drug Administration (FDA) for the treatment of non-small-cell lung cancer (NSCLC). Bexarotene is approved by the FDA for the treatment of cutaneous T-cell lymphoma. This combination of drugs is experimental.

DETAILED DESCRIPTION:
This is a single institution open label phase II trial. Consecutive, eligible patients presenting with the diagnosis of advanced NSCLC are to be enrolled in this study. All eligible patients will receive continuous daily oral erlotinib 150 mg (Tarceva™) with daily bexarotene oral capsules 400 mg/m2 (Targretin®). The two agents will be taken at the same time. We anticipate the maximum accrual of 40 patients to this trial.

Patients will be evaluated by history, physical examination, and laboratory assessment every 4 weeks. Radiographic disease assessments by chest radiograph will be obtained every 4 weeks and computer tomography every 8 weeks or longer if clinically indicated. Whole body PET scan will be obtained at 10 days and 8 weeks. All radiographic studies will be sent to Medical Metrix Solutions (MMS) for an independent radiographic review of tumor response.

ELIGIBILITY:
Inclusion Criteria:

* Advanced NSCLC
* Prior chemotherapy or radiotherapy is allowed.

Exclusion Criteria:

* Hepatic or renal dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-08; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin H Dragnev, MD, Principal Investigator — Norris Cotton Cancer Center
Locations (2):
- United States (2):
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - Mount Sinai School of Medicine, New York, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Erlotinib + Bexarotene: All eligible patients will receive continuous daily oral erlotinib 150mg with daily bexarotene oral capsules 400mg.
  erlotinib and bexarotene: Daily Erlotinib 150mg and daily bexarotene oral capsules 400mg.
Period: Overall Study
Arm/Group | Single Arm Erlotinib + Bexarotene
Started | 42
Completed | 19
Not Completed | 23
Not completed — Death | 4
Not completed — Adverse Event | 5
Not completed — Physician Decision | 14

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Erlotinib + Bexarotene
Number analyzed (Participants) | 42
Age, Continuous [Median (Full Range); unit: years] | 67 [46 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 42
Disease Stage IV [Count of Participants; unit: Participants] — The clinical stage of disease for participants will be Stage IV (Stage 4) disease. Staging is based on different characteristics of the cancer diagnosis that determine how advanced the cancer is.
  Participants | 42
Histopathology [Number; unit: participants] — Includes multiple histopathology types (adenocarcinoma and brochioloalveolar type).
  participants
    Adenocarcinomas | 28
    Bronchioloalveolar type | 5
    Squamous cell carcinoma | 2
    Non-small cell carcinomas not otherwise specified | 10
Prior anti-EGFR therapy [Count of Participants; unit: Participants]
  Received prior anti-EGFR therapy | 9
  Did not receive prior anti-EGFR therapy | 33
Number of prior chemotherapies [Median (Full Range); unit: chemotherapies] | 2 [0 to 5]
Smoking status [Count of Participants; unit: Participants]
  Never smoker | 7
  Current smoker | 6
  Former smoker | 29

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Response Rates
Description: Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Erlotinib + Bexarotene
Number analyzed (Participants) | 19
Participants | 19

2. Secondary Outcome: Correlation of Early PET Responses With Objective Radiographic Responses.
Description: PET response is assessed based on the guidelines of the European Organization for Research and Treatment of Cancer (EORTC) PET Study Group (Eur J Cancer 1999; 35(13):1773-82). PET response refers to the presence and measurement of the most current PET scan imaging when compared to baseline imaging. The amount of reduction in the disease from baseline to current imaging determines the extent to which the cancer has responded to treatment. Radiographic response is per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: Through study completion, an average of 1 year
Population: Number of participants analyzed is reported per achieved disease response noted in individual rows.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Erlotinib + Bexarotene
Number analyzed (Participants) | 14
Participants
  Computed tomography complete response: number analyzed (Participants) | 1
  Computed tomography complete response: Early PET metabolic response | 1
  Computed tomography complete response: Early PET metabolic progression | 0
  Computed tomography complete response: Early PET stable disease | 0
  Computed tomography complete response: Early PET progression | 0
  Computed tomography partial response: number analyzed (Participants) | 1
  Computed tomography partial response: Early PET metabolic response | 0
  Computed tomography partial response: Early PET metabolic progression | 1
  Computed tomography partial response: Early PET stable disease | 0
  Computed tomography partial response: Early PET progression | 0
  Computed tomography stable disease: number analyzed (Participants) | 2
  Computed tomography stable disease: Early PET metabolic response | 0
  Computed tomography stable disease: Early PET metabolic progression | 0
  Computed tomography stable disease: Early PET stable disease | 1
  Computed tomography stable disease: Early PET progression | 1
  Computed tomography disease progression: number analyzed (Participants) | 10
  Computed tomography disease progression: Early PET metabolic response | 0
  Computed tomography disease progression: Early PET metabolic progression | 0
  Computed tomography disease progression: Early PET stable disease | 5
  Computed tomography disease progression: Early PET progression | 5

3. Secondary Outcome: Progression-free Survival and Overall Survival
Time Frame: Through study completion, an average of 1 year
Measure: Median (Full Range); unit: Weeks
Arm/Group | Single Arm Erlotinib + Bexarotene
Number analyzed (Participants) | 40
Weeks
  Time to progression | 7 [1 to 274]
  Overall survival | 22 [1 to 274]

4. Secondary Outcome: Evaluation of EGFR Mutations in Tumor Biopsies and Correlation of EGFR Mutations With Objective Radiographic Responses.
Time Frame: Through study completion, an average of 1 year
Population: Three patients had biopsies evaluated for EGFR mutations.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Erlotinib + Bexarotene
Number analyzed (Participants) | 3
Participants
  Complete Response (CR) in EGFR Wild-Type | 0
  Partial Response in EGFR Wild-Type | 2
  CR in Activating EGFR mutation at exon 21 | 1
  PR in Activating EGFR mutation at exon 21 | 0

ADVERSE EVENTS:
Arm/Group | Single Arm Erlotinib + Bexarotene
All-Cause Mortality (participants affected / at risk) | 4/42
Serious Adverse Events (participants affected / at risk) | 30/42
Other Adverse Events (participants affected / at risk) | 14/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Erlotinib + Bexarotene (N=42)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Chest pain (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 2
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 3
Anxiety Disorder (Psychiatric disorders) | 1
Post-obstructive Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2
Bacterial pneumonia (Infections and infestations) | 1
Mental status changes (Psychiatric disorders) | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pain (Musculoskeletal and connective tissue disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Declining respiratory status (Respiratory, thoracic and mediastinal disorders) | 1
Acute renal failure (Renal and urinary disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm Erlotinib + Bexarotene (N=42)
Hallucinations (Psychiatric disorders) | 1
Fatigue (General disorders) | 3
INR increased (Investigations) | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 5 (16)
Activated partial thromboplastin time prolonged (Investigations) | 1
Increased white blood cell count (Blood and lymphatic system disorders) | 1
Investigations - Other, elevated granulocytes (Investigations) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Proximal muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 1
Cholesterol high (Investigations) | 1
Mouth sores (Gastrointestinal disorders) | 1
Arm pain (Musculoskeletal and connective tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes